CLINICAL TRIAL: NCT04107259
Title: Circulating IRAPe, Irisin and IL-34 in Relation to Insulin Resistance in Patients With Type 2 Diabetes
Brief Title: IRAPe, Irisin and IL-34 in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Other Study IDs: IRAPe, Irisin and IL-34
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; IL-34; Irisin; IRAPe; Visfatin; Insulin resistance; HOMA-IR
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with diabetes: 60 newly diagnosed type 2 diabetes
  Interventions: Diagnostic Test: Blood sample
- Control: 60 non-diabetic control subjects
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Ten ml of venous blood was collected from all participants in the early morning after an overnight 12 hour fast by venipuncture of the antecubital vein into sterile tubes. Plasma and sera were separated immediately and were stored at -70 C until biochemical analyses.

SUMMARY:
Aim: This study aimed to evaluate the role of extracellular part of insulin regulated aminopeptidase (IRAPe), IL-34, Irisin, and Visfatin in the development of insulin resistance in patients with type 2 diabetes mellitus.

Methods: parallel study enrolled 60 non-diabetic control subjects and 60 newly-diagnosed type 2 diabetics, matched for age, body mass index and sex ratio.

DETAILED DESCRIPTION:
Aim: This study aimed to evaluate the role of extracellular part of insulin regulated aminopeptidase (IRAPe), IL-34, Irisin, and Visfatin in the development of insulin resistance in patients with type 2 diabetes mellitus.

Methods: parallel study enrolled 60 non-diabetic control subjects and 60 newly-diagnosed type 2 diabetics, matched for age, body mass index and sex ratio. Anthropometric parameters, blood glucose, fasting plasma insulin, insulin resistance index (HOMA-IR), IL34, Irisin, IRAPe, Visfatin and glycated hemoglobin were assessed.

Conclusion: IL-34 and Visfatin levels were significantly increased, while both Irisin and IRAPe levels were significantly decreased in patients with type 2 diabetes. Theses aforementioned parameters were significantly correlated with insulin resistance. These findings indicate that, IL-34, Irisin and IRAPe may play a vital role in T2DM and in diabetes associated insulin resistance. Additionally, the investigator's findings proposed that, IRAPe may be a useful and direct marker for detection of insulin resistance state.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes and non-diabetic control subjects from 35 to 65 years old were enrolled in this study.

Exclusion Criteria:

* individuals with inflammatory diseases, Cushing's syndrome, thyroid disorders, infectious diseases, cancers, hepatic diseases and renal impairment. Subjects on insulin or other medications that could affect glucose metabolism or pro-inflammatory cytokines assessment (Glucocorticoids, beta-Adrenergic agonists, Thiazides, etc.....) were also excluded from study

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus were diagnosed according to the criteria of the World Health Organization. All individuals included in this study were adult Middle-Eastern Egyptian citizens and were subjected to full medical history and physical examination by hospital physicians.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose (FBG) levels | three months
  were assayed using glucose oxidase method.
Fasting plasma insulin (FPI) | three months
  was assayed using Enzyme-Linked Immunosorbent Assay kits i.e ELISA
HOMA-IR index | three months
  HOMA-IR index which is defined as fasting insulin (μIU/ml) times fasting glucose (mg/L) divided by 405 if fasting blood glucose is expressed in mass units (mg/dl).
plasma IL-34 | Three months
  human plasma IL-34 was assayed using sandwich enzyme immunoassay technique
serum visfatin | Three Months
  serum visfatin concentrations enzyme- immunoassay kit
IRAPe | Three months
  extracellular part of insulin regulated aminopeptidase (IRAPe) level was determined using sandwich enzyme immunoassay technique

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mostafa, Ass Prof., Study Chair — Tanta University
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

REFERENCES:
- [Result] Chang EJ, Lee SK, Song YS, Jang YJ, Park HS, Hong JP, Ko AR, Kim DY, Kim JH, Lee YJ, Heo YS. IL-34 is associated with obesity, chronic inflammation, and insulin resistance. J Clin Endocrinol Metab. 2014 Jul;99(7):E1263-71. doi: 10.1210/jc.2013-4409. Epub 2014 Apr 8. PMID 24712570
- [Result] Sesti G, Andreozzi F, Fiorentino TV, Mannino GC, Sciacqua A, Marini MA, Perticone F. High circulating irisin levels are associated with insulin resistance and vascular atherosclerosis in a cohort of nondiabetic adult subjects. Acta Diabetol. 2014 Oct;51(5):705-13. doi: 10.1007/s00592-014-0576-0. Epub 2014 Mar 12. PMID 24619655
- [Derived] Mostafa TM, El-Gharbawy NM, Werida RH. Circulating IRAPe, Irisin, and IL-34 in Relation to Insulin Resistance in Patients With Type 2 Diabetes. Clin Ther. 2021 Jul;43(7):e230-e240. doi: 10.1016/j.clinthera.2021.05.003. Epub 2021 Jun 5. PMID 34103176